CLINICAL TRIAL: NCT01062282
Title: VENIS - Prospective Observational Study of Ventavis® Inhalation Therapy in the Treatment of Patients With Pulmonary Arterial Hypertension
Brief Title: Hypertension Study of Ventavis® Inhalation Therapy in the Treatment of Patients With Pulmonary Arterial Hypertension (VENIS)
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer Korea LTD
Other Study IDs: 14184; VENIS; VE0610KR
Record Dates: First submitted 2009-08-20; First posted 2010-02-04 (Estimated); Last update posted 2011-04-04 (Estimated); Status verified 2011-04

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Iloprost

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Iloprost (Ventavis BAYQ6256)

INTERVENTIONS:
Drug: Iloprost (Ventavis BAYQ6256) — Patients with pulmonary arterial hypertension, classified as New York Heart Association functional class III or IV where the treating physician has chosen Ventavis as a suitable treatment prior to inclusion into this non-interventional study. Patients should not have received prior treatment with Ventavis

SUMMARY:
The purpose of this study is to gain information on safety and efficacy from Korean patients who starting Ventavis treatment by observational method.

ELIGIBILITY:
Inclusion Criteria:

* The treating physician has chosen Ventavis as a suitable treatment for the patient
* Patient with PH and classified as NYHA functional class III or IV and WHO group 1

Exclusion Criteria:

* Any condition that prevents participation in the study, including pregnancy and other contraindications for Ventavis treatment (as listed in the current Ventavis patient package insert).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary hypertension in Korea
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2006-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable is 6-minute walking distance | At baseline and month 1,3,6 for an observational period of 6 months

SECONDARY OUTCOMES:
New York Heart Association functional class | Baseline, month 1,3,6
PH-related symptoms and change of concomitant medication | Baseline, month 1,3,6
Hemodynamic parameters | If applicable ( at any time during Ventavis treatment)
Adverse Event collection | If applicable (during the study period)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, South Korea